CLINICAL TRIAL: NCT01870895
Title: A Double-blind, Parallel-group, Comparative Study in Female Patients With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: A Study to Assess the Efficacy and Safety of YM060 in Female Patients With Diarrhea-predominant Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060-CL-702
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
Keywords: YM060; Ramosetron; Diarrhea-predominant Irritable Bowel Syndrome
MeSH Terms: interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- YM060 group (Experimental)
  Interventions: Drug: YM060
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YM060 — oral
  Other Names: ramosetron,; Irribow
  Arms: YM060 group
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
To demonstrate the superiority of YM060 to a placebo in global assessment of relief of overall IBS symptoms and stool form normalization, and to evaluate safety in female patients with diarrhea-predominant irritable bowel syndrome (D-IBS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients satisfying the Rome III Diagnostic Criteria
2. Patients whose ≥25% of stools were loose or watery and <25% of them were hard or lumpy stools
3. Patients who have abdominal pain or discomfort
4. Patients in whom after occurrence of IBS symptoms the following tests were conducted and in whom no organic changes were observed Pancolonoscopy or contrast enema

Exclusion Criteria:

1. Patients with a history of surgical resection of the stomach, gallbladder, small intestine or large intestine
2. Patients with a history or current evidence of inflammatory bowel disease
3. Patients with a history or current evidence of colitis ischemic
4. Patients with concurrent infectious enteritis
5. Patients with concurrent hyperthyroidism or hypothyroidism
6. Patients with concurrent active peptic ulcer
7. Patients with other concurrent disease that may affect the digestive tract passage or large intestinal function or that is likely to interfere with proper assessment of IBS abdominal pain/discomfort

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 577 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Monthly responder rate of global assessment of relief of overall IBS symptoms at final point | Up to 12 weeks
Monthly responder rate of stool form normalization at final point | Up to 12 weeks

SECONDARY OUTCOMES:
Monthly responder rate of global assessment of relief of abdominal pain/discomfort | Up to 12 weeks
Monthly responder rate of global assessment of improvement of abnormal bowel habits | Up to 12 weeks
Change in weekly average scores of severity of abdominal pain/discomfort | Up to 12 weeks
Change in weekly average scores of stool form | Up to 12 weeks
Safety assessment of YM060 | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu

REFERENCES:
- [Derived] Fukudo S, Kinoshita Y, Okumura T, Ida M, Akiho H, Nakashima Y, Nishida A, Haruma K. Ramosetron Reduces Symptoms of Irritable Bowel Syndrome With Diarrhea and Improves Quality of Life in Women. Gastroenterology. 2016 Feb;150(2):358-66.e8. doi: 10.1053/j.gastro.2015.10.047. Epub 2015 Nov 6. PMID 26551550
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=060-CL-702